CLINICAL TRIAL: NCT00189293
Title: Multicenter, Randomised, Double-blind, Vehicle-controlled Study Comparing Recurrence Rate Following Imiquimod 5% Cream or Vehicle 3 Times Per Week for 4 Weeks Prior to Ablative Therapy in Subjects Suffering From External Ano-Genital Warts
Brief Title: Study of Imiquimod Cream Prior to Ablative Therapy in External Ano-Genital Warts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Responsible Party: Joachim Maus, MD, Director Clinical Development, Meda Pharma GmbH & Co. KG
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1526-IMIQ; 2004-004654-19 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2008-09

CONDITIONS: Genital Warts
Keywords: External Ano-Genital Warts; Ablative Therapy; Aldara
MeSH Terms: conditions — Condylomata Acuminata | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Imiquimod 5% cream
  Interventions: Drug: Imiquimod
- 2 (Other): vehicle cream
  Interventions: Other: vehicle cream

INTERVENTIONS:
Drug: Imiquimod — Imiquimod 5% cream three times per week for 4 weeks (1 sachet)
  1 or 2 sachet(s)
  Arms: 1
Other: vehicle cream — vehicle cream three times per week for 4 weeks (1 sachet)
  1 or 2 sachet(s)
  Arms: 2

SUMMARY:
The purpose of this study is to compare the recurrence rate following total clearance of external genital warts (EGWs) when clearance has been obtained by imiquimod (3 applications per week for 4 weeks) followed by ablative therapy (laser or electrocautery therapy) with that from just ablative therapy treatment alone.

DETAILED DESCRIPTION:
To compare the recurrence rate 24 weeks after ablative therapy in subjects with external genital warts trated with imiquimod, 3 applications per week for 4 weeks followed by ablative therapy versus vehicle, 3 applications per week for 4 weeks followed by ablative therapy. A recurrence is defined as the investoigator-assessed occurrence of lesion(s) within the baseline area cleared by the treatment: imiquimod/vehicle then ablative therapy (either the initial ablative therápy session (A0), or if required for complete clearance of baseline lesions, a second ablative therapy session (A2).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with at least 1 visible genital or perianal wart
* Total wart area 1 to 40 square centimeters.

Exclusion Criteria:

* Pregnant or lactating women
* Known other sexually transmitted disease
* Evidence of a clinically significant immunodeficiency
* Evidence of unstable cardiovascular, pulmonary, hematological, hepatic, renal, endocrine, collagen vascular, neurological or gastrointestinal abnormality or disease.
* Treatment within the 4 weeks prior to the Randomization Visit with any of the following systemic or topical treatments: interferons, interferon inducers, immunomodulators, immunosuppressive drugs, antiviral drugs (except for systemic acyclovir, valacyclovir and famciclovir), cytotoxic drugs, investigational drugs, or any drugs known to have major organ toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
recuurence rate 24 weeks after ablative therapy | 24 weeks

SECONDARY OUTCOMES:
Time to recurrence
Recurrence rate at 4 and 12 weeks post ablation | 4 and 12 weeks
Reduction of EGW area | 4 and 12 weeks
Healing and cosmetic outcome | 4, 12 and 24 weeks
Local and general tolerability
Percent of complete clearance after initial topical treatment | up to 6 weeks after initial topical treatment
Occurrence of new lesions

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Boselli, MD, Principal Investigator — Unità di Ginecologia Preventiva e Oncologica Università di Modena e Reggio Emilia
Locations (12):
- Italy (12):
  - Clinica Ostetrica e Ginecologica Università Politecnica delle Marche, Ancona
  - Struttura Complessa di Ostetricia e Ginecologia Ospedale Cardinal Massaia, Asti
  - Unità Operativa di Ginecologia Oncologica, RCCS Ospedale Oncologico, Bari
  - Servizio Autonomo di Diagnosi Precoce dei Tumori Ginecologici Ospedale Vittorio Emanuele, Catania
  - Clinica Ostetrica Ginecologica, Ospedale Careggi, Florence
  - Struttura Complessa Oncologia Chirurgica C Istituto Scientifico dei Tumori IST, Genova
  - Servizio di Ginecologia Preventiva, Istituti Clinici di Perfezionamento, Milan
  - Clinica Ostetrica Ginecologica Azienda Ospedaliera L. Sacco, Milan
  - Unità di Ginecologia Preventiva e Oncologica Università di Modena e Reggio Emilia, Modena
  - Unità Operativa di Ginecologia Oncologica, Ospedale Oncologico M. Ascoli, Palermo
  - Ostetricia e Ginecologia, Ospedale S. Maria delle Grazie, Pozzuoli
  - Ambulatorio di Colposcopia e Patologia Cervico-Vaginale, Università Cattolica del Sacro Cuore, Roma